CLINICAL TRIAL: NCT04933734
Title: Turkish Cultural Adaptation, Validity and Reliability of the "Physical Activity-Specific Rumination Scale for Children"
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assist. Prof., Istanbul University - Cerrahpasa
Other Study IDs: NArman
Record Dates: First submitted 2021-06-13; First posted 2021-06-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Children, Only; Physical Activity; Rumination
Keywords: Rumination; Children; Intrinsic barriers
MeSH Terms: conditions — Motor Activity; Rumination Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anxiety that turns into an over-generalized and repetitive form is called rumination. When the literature was reviewed, rumination was found to be associated with depression and anxiety, but its applicability to physical activity (PA) behaviors has been largely overlooked. Only a few studies have examined the relationship between rumination and PA behaviors. The study was designed with the aim of determining the Turkish cultural adaptation, validity and reliability of the "Physical Activity-Specific Rumination Scale for Children (PARS-C)" questionnaire developed for children in England in order to determine the intrinsic factors affecting participation in PA.

DETAILED DESCRIPTION:
Rumination is the individual's persistent thinking about the negative mood, symptoms, possible causes and consequences; however, it is defined as not taking action to solve the problem. When the literature was reviewed, it was found that rumination in children was associated with depression and anxiety, but information about its applicability to PA behaviors is limited. Only a few studies have examined the relationship between rumination and PA behaviors. The importance of identifying the intrinsic barriers and facilitators that affect participation in FA in children is frequently emphasized. For this purpose, the "Physical Activity-Specific Rumination Scale for Children (PARS-C)" scale, which evaluates the relationship between FA and rumination, was developed for the first time in England. It has been reported that PARS-C is a useful tool to evaluate children's PA-specific rumination tendencies and to improve our understanding of the role of rumination in PA behavior, but its applicability to other cultures requires further research. The present study was designed with the aim of determining the Turkish cultural adaptation, validity and reliability of the "Physical Activity-Specific Rumination Scale for Children (PARS-C)" questionnaire. To evaluate the validity, The Physical Activity Questionnaire for Older Children (PAQ-C) and Motivation Scale For Participation In Physical Activity (MSPPA) will be applied. To evaluate reliability, the Turkish form of PARS-C will be applied again after 7 days. All forms will be sent to children in google forms format.

It is planned to include 500 children in this study. Factor analysis methods will be used in the analysis of the factor structure of the scale, correlation analyzes (Pearson and Spearman coefficients) will be used in the analysis of validity and test-retest reliability. Cronbach's alpha analysis will be used in the reliability analysis. The study will be the first to reveal the relationship between FA behavior and rumination in Turkish children. The results will contribute to the determination of FA barriers in Turkish children.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Not having any diagnosed disease
* 8-14 ages
* Have reading and writing skills
* Studying in primary or secondary school level
* Residing in Turkey
* To have the cognitive skills to understand and answer the questions in the questionnaires

Exclusion Criteria:

* Having a vision or hearing problem
* Have a diagnosed chronic cardiac, neurological, or rheumatic disease

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 8-14 years at primary or secondary school level who meet the inclusion criteria will be included in our study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
"Physical Activity-Specific Rumination Scale for Children (PARS-C)" (Time Frame: Change from baseline to 7 day) | Time Frame: Change from baseline to 7 day
  It was developed by Ling et al. It evaluates rumination tendencies related to physical activity in children. Consisting of 10 items, PARS-C is a 3-point Likert type scale. In our study, rumination tendencies of children related to FA will be evaluated with PARS-C.
The Physical Activity Questionnaire for Older Children ( PAQ-C) (Baseline) | Baseline
  It was developed by Kowalski et al. The PAQ-C is a seven-day self-report scale designed to assess moderate-to-vigorous physical activity in children aged 8-14 years. This questionnaire contains nine items and examines the physical activities performed by the student in the last seven days and the frequency of these activities. In this study children's physical activity levels will be evaluated with the PAQ-C.
Motivation Scale For Participation In Physical Activity (MSPPA) (Baseline) | Baseline
  MSPPA was developed by Tekkursun Demir and Cicioglu. It was developed to assess children's motivation to participate in physical activity. The scale, which consists of 16 items, is in the 5-point Likert type. In our study, children's motivations about physical activity will be evaluated with MSPPA.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Asst. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No